CLINICAL TRIAL: NCT03496870
Title: A Phase 1, Open-Label Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Repeated Doses of Opicapone, and Effect on Levodopa Pharmacokinetics in Subjects With Parkinson's Disease
Brief Title: A Study of the Pharmacokinetics, Pharmacodynamics, and Safety of Opicapone in Subjects With Parkinson's Disease Taking Levodopa.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-OPC-1706
Record Dates: First submitted 2018-03-01; First posted 2018-04-12 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Opicapone once daily with Carbidopa/Levodopa (Experimental): Opicapone administered once daily for 14 days; carbidopa/levodopa administered at set frequency on Study Days 1, 2 & 15
  Interventions: Drug: Opicapone; Drug: Carbidopa Levodopa

INTERVENTIONS:
Drug: Opicapone — catechol-O-methyltransferase (COMT) inhibitor
  Other Names: BIA 9-1067
Drug: Carbidopa Levodopa — Levodopa: dopamine precursor Carbidopa: DOPA decarboxylase inhibitor
  Other Names: Sinemet

SUMMARY:
This is a phase 1, open-label study to assess the pharmacokinetics, pharmacodynamics, safety, and tolerability of opicapone when administered orally once daily for 14 days as adjunctive therapy to carbidopa/levodopa in subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of idiopathic Parkinson's Disease (PD) for at least 3 years with clear improvement with levodopa treatment
2. Be at a stable dose of maintenance medication(s) for PD, including stable doses of CD/LD
3. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study
4. Have a body mass index (BMI) of 18 to 40 kg/m2
5. Have a modified Hoehn and Yahr stage of ≤4 in the OFF state
6. Be able to tolerate an overnight period of 12 hours without CD/LD
7. Be in good general health and expected to complete the clinical study as designed

Exclusion Criteria:

1. Are currently pregnant or breastfeeding
2. More than 2 alcoholic beverages daily or more than 14 alcoholic beverages weekly within 7 days of Day -1 or consume any alcohol within 48 hours of Day -1.
3. Have motor fluctuations during the day (ie, effect of levodopa "wearing off" or having unpredictable "off" periods), or severe or intolerable levodopa-induced dyskinesia
4. Have had previous exposure to opicapone, or have an allergy, hypersensitivity, or intolerance to opicapone or other COMT inhibitor.
5. Have a history of a medical condition or surgical procedure that might interfere with absorption or metabolism.
6. Have a known history of neuroleptic malignant syndrome
7. Have an unstable medical condition or chronic disease
8. Have taken certain prohibited medications within 28 days of Day -1.
9. Have a known or suspected diagnosis of AIDS, or have tested seropositive for HIV
10. Have hepatitis A or B
11. Have a significant risk of suicidal or violent behavior

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic evaluation of opicapone and its metabolites: area under the curve (AUC 0-24) | up to 19 days
  Area under the plasma concentration versus time curve from 0 to 24 hours for analytes with quantifiable concentrations at 24 hours postdose
Pharmacokinetic evaluation of opicapone and its metabolites: area under the curve (AUC 0-tlast) | up to 19 days
  Area under the plasma concentration versus time curve from 0 hour to the time of the last measurable concentration for analytes below the limit of quantification at 24 hours postdose
Pharmacokinetic evaluation of opicapone and its metabolites: Maximum plasma concentration (Cmax) | up to 19 days
  Maximum plasma concentration
Pharmacokinetic evaluation of opicapone and its metabolites: Time to maximum plasma concentration (tmax) | up to 19 days
  Time to maximum plasma concentration
Pharmacokinetic evaluation of levodopa following administration of opicapone: area under the curve (AUC 0-tlast) | up to 15 days
  Area under the plasma concentration versus time curve from 0 hours to time before next levodopa dose
Pharmacokinetic evaluation of levodopa following administration of opicapone: maximum plasma concentration (cmax) | up to 15 days
  Maximum plasma concentration

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | up to 19 days
  Number of participants with reported adverse events after study treatment.
Pharmacodynamic evaluation of opicapone on S-COMT activity | up to 19 days
  Maximum inhibition of S-COMT activity.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Chief Medical Officer
Locations (3):
- United States (3):
  - Neurocrine Clinical Site, Glendale, California
  - Neurocrine Clinical Site, Long Beach, California
  - Neurocrine Clinical Site, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: No